CLINICAL TRIAL: NCT06015711
Title: The Effect of Preoperative Maxigesic® Administration on Analgesic Nociception Index (ANI) Guided Remifentanil Administration
Brief Title: The Effect of Preoperative Maxigesic® on Intraoperative Remifentanil Requirement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, In-kyong Yi, Assitant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: AJOUIRB-IV-2023-400
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Opioid Use

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maxigesic group (Experimental): Administration of Maxigesic before surgery start.
  Interventions: Drug: Maxigesic administration
- Control group (No Intervention): Administration of normal saline before surgery start.

INTERVENTIONS:
Drug: Maxigesic administration — Preoperative Maxigesic IV administration
  Other Names: Preoperative Maxigesic administration
  Arms: Maxigesic group

SUMMARY:
Maxigesic is combined intravenous analgesic of ibuprofen and acetaminphen. The purpose of this study is investigate weather preoperative Maxigesic administration can reduce intraoperative remifentanil requirement.

DETAILED DESCRIPTION:
Remifentanil is an ultra-short-acting opioid that is useful during surgery because of its fast onset and recovery. However, because of this profile, it is known that the use of high doses of remifentanil during surgery paradoxically increases postoperative pain. It has been reported that intraoperative remifentanil use resulted in higher pain scores 2 hours after surgery compared to intraoperative dexmedetomidine, and that the incidence of hypotension, tremor, and postoperative nausea and vomiting were higher in the remifentanil group. Therefore, minimizing the use of remifentanil during surgery is clinically meaningful.

Nonsteroidal anti-inflammatory drugs (NSAIDs) play an important role in multimodal analgesia, and are known to reduce the use of opioids when used together with opioids in postoperative pain [3]. It has also been reported that preoperative administration of ibuprofen reduces postoperative opioid use. Administration of acetaminophen has also been reported to reduce opioid usage. However, there is no study on whether the administration of these NSAIDs and acetaminophen reduces the opioid requirement used during surgery, not after surgery.

The Analgesia nociception index (ANI, MDoloris medical system, France) was developed to measure real-time nociception in patients undergoing surgery under general anesthesia. This index measures parasympathetic nerve activity based on heart rate variability. It is known to be superior in detecting nociceptive stimuli rather than judging only by existing pulse rate and blood pressure. In addition, since information is provided as an objectified numerical value, analgesic drugs can be adjusted during surgery based on this information. This helps to provide an appropriate amount of opioids during surgery when needed, and can prevent overdose. A previous study reported that when ANI-guided remifentanil infusion was performed, the amount of remifentanil used was reduced compared to conventional control of remifentanil only with blood pressure and pulse rate.

Maxigesic® is a combination of acetaminophen and ibuprofen, and is a drug that rapidly relieves various types of pain. It is known to be more effective in relieving postoperative pain than single acetaminophen or ibuprofen. The hypothesis of this study is that administration of Maxigesic®, a combination of acetaminophen and NSAIDs, reduces intraoperative remifentanil requirement. This study aims to investigate whether preoperative Maxigesic® administration can reduce intraoperative remifentanil requirements by performing ANI-guided remifentanil infusion for objective control of remifentanil administration.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (19-60 years old) with ASA physical status 1, 2, 3
* Scheduled surgery under general anesthesia

Exclusion Criteria:

* The patient does not conset
* Pregnancy
* hepatic disorder
* Renal disorder
* Asthma
* Hypersensitivity to the NSAIDs or acetaminophen
* Patients receiving chronic pain therapy
* Drug dependence
* Patients taking psychiatric drugs
* Alcoholics
* History of gastrointestinal ulcer or bleeding

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Remifentanil requirement | 3 hours, from incision to skin closure
  Intraoperative remifentanil requirement

SECONDARY OUTCOMES:
postoperative analgesic requirement | 1 hour, while in the recovery room
  postoperative fentanyl requirement

CONTACTS AND LOCATIONS:
Overall Officials: In Kyong Yi, MD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou university school of medicine, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No
In case of individual reasonable request to PI